CLINICAL TRIAL: NCT06400511
Title: A Randomized, Double-Masked, Vehicle-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Pimecrolimus 0.3% Ophthalmic Ointment (MR-139), in Subjects With Blepharitis
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Pimecrolimus 0.3% Ophthalmic Ointment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Famy Life Sciences, a Viatris Company (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCLS-OMZ-3001
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pimecrolimus 0.3% Ophthalmic Ointment (Active Comparator): Study Drug
  Interventions: Drug: Pimecrolimus 0.3% Ophthalmic Ointment
- Placebo Ophthalmic Ointment (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Ophthalmic Ointment

INTERVENTIONS:
Drug: Pimecrolimus 0.3% Ophthalmic Ointment — Pimecrolimus 0.3% Ophthalmic Ointment will be applied twice a day to both eyelid margins.
  Arms: Pimecrolimus 0.3% Ophthalmic Ointment
Drug: Placebo Ophthalmic Ointment — Placebo will be applied twice a day to both eyelid margins.
  Arms: Placebo Ophthalmic Ointment

SUMMARY:
The objective of this study is to determine the efficacy and safety of Pimecrolimus 0.3% (MR-139) Ophthalmic Ointment.

DETAILED DESCRIPTION:
The study is designed to evaluate Pimecrolimus 0.3% Ophthalmic Ointment in subjects with blepharitis to complete resolution (score = 0 on grading scale of 0-4) for eyelid debris after BID use at Week 6 in the Study Eye.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 2 years of age or older at Visit 1, with a diagnosis of blepharitis confirmed by the investigator.
2. Subjects under 18 must able to be examined at the slit lamp (handheld) without systemic anesthesia.
3. A self-reported history of at least 1 previous episode of blepharitis.
4. Adult subjects have provided verbal and written informed consent. For subjects under 16 years of age, a parent or legal guardian of each subject must provide written informed consent and sign the HIPAA form (or equivalent, if applicable), approved by the appropriate Institutional Review Board (IRB)/Ethical Committee (EC). Whenever practical and appropriate per local requirements, a child's assent should also be sought before inclusion into the study.
5. Subjects who have not responded adequately to lid hygiene in the past (self-reported).
6. Have a Corrected Distance Visual Acuity (CDVA) greater than or equal to 0.7 logMar in each eye, assessed with the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. Subjects may be refracted if needed.
7. Subjects must be able to comply with the requirements of the protocol including the ability to self-administer or receive topical treatment twice a day to their eyelid margins.
8. Be literate and able to complete questionnaires independently, or in the case of pediatric patients, can comprehend the questionnaires with the help of a parent/guardian or interviewer.
9. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at Visit 1 and must be willing to use an adequate method of contraception throughout the study and 30 days from the last application of the study treatment.

Exclusion Criteria:

1. Subjects who have received a COVID vaccination or recovered from COVID-19 symptoms less than 1 week prior to baseline visit.
2. Subjects with a history of, or active herpetic or neurotrophic keratitis.
3. Subjects who, in the opinion of the investigator, have abnormal eyelid anatomy (other than due to blepharitis) that might adversely affect clinical signs and symptoms, including but not limited to lagophthalmos, malposition of the eyelid or tumor(s) of the eyelid or eyelid margin.
4. Subjects who have received other treatments for blepharitis within 30 days of Visit 1.
5. Subjects with known hypersensitivity to study medications, or to any diagnostic agents to be used in the study.
6. Subjects who are currently enrolled in an investigational drug or device study or have used an investigational drug or device within the 30 days prior to the baseline visit and during the treatment period.
7. Subjects who, in the opinion of the investigator, would be unable to adhere to the study protocol.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of Study Drug | 6 weeks
  Complete Resolution (score =0 on grading scale 0-4) of eyelid debris. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Ocular Discomfort Score | 6 weeks
  Proportion with at least 50% reduction from baseline in ODS at Week 6. Ocular discomfort is assessed by visual analog scale on a scale from 0-100 where 0 indicates no discomfort and 100 indicates maximum. A higher score indicates a worse outcome.
Collarettes | 6 weeks
  Proportion of complete resolution for collarettes (score =0 on grading scale 0-4) at Week 6. A higher score indicates a worse outcome.
Eyelid Redness | 6 weeks
  Proportion of complete resolution (score =0 on grading scale 0-4) for eyelid redness (erythema) at Week 6. A higher score indicates a worse outcome.
Ocular Discomfort Score | 6 weeks
  The mean change from baseline in ODS at Week 6. Ocular discomfort is assessed by visual analog scale on a scale from 0-100 where 0 indicates no discomfort and 100 indicates maximum. A higher score indicates a worse outcome.
Blepharitis Symptom Measurement | 6 weeks
  Proportion of complete resolution (score =0 on grading scale of 0-3) for the Eye Irritation Symptom on the BLISS at Week 6. A higher score indicates a worse outcome.
Eyelid Meibum Character | 6 weeks
  Proportion of complete resolution (score = 0 on grading scale 0-24 for upper lid; 0-15 for lower lid) for eyelid meibum character at Week 6. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Macsai, MD, Study Director — Viatris Eye Care Division
Locations (29):
- United States (29):
  - Clinical Investigative Site, Pheonix, Arizona
  - Clinical Investigator Site, Garden Grove, California
  - Clinical Investigator Site, Glendale, California
  - Clinical Investigator Site, Inglewood, California
  - Clinical Investigator Site, Newport Beach, California
  - Clinical Investigator Site, Petaluma, California
  - Clinical Investigator Site, Rancho Cordova, California
  - Clinical Investigator Site, Aurora, Colorado
  - Clinical Investigator Site, Crystal River, Florida
  - Clinical Investigator Site, Largo, Florida
  - Clinical Investigator Site, Tampa, Florida
  - Clinical Investigator Site, Atlanta, Georgia
  - Clinical Investigator Site, Morrow, Georgia
  - Clinical Investigator Site, Pittsburg, Kansas
  - Clinical Investigator Site, Louisville, Kentucky
  - Clinical Investigator Site, Havre de Grace, Maryland
  - Clinical Investigator Site, Medina, Minnesota
  - Clinical Investigator Site, Kansas City, Missouri
  - Investigative Site, St Louis, Missouri
  - Clinical Investigator Site, Washington, Missouri
  - Clinical Investigator Site, Garner, North Carolina
  - Clinical Investigator Site, Cincinnati, Ohio
  - Clinical Investigator Site, Cranberry Township, Pennsylvania
  - Clinical Investigator Site, Smyrna, Tennessee
  - Clinical Investigator Site, Austin, Texas
  - Clinical Investigator Site, Lakeway, Texas
  - Clinical Investigator Site, San Antonio, Texas
  - Clinical Investigator Site, Clinton, Utah
  - Clinical Investigator Site, Lynchburg, Virginia